CLINICAL TRIAL: NCT05521685
Title: Impact of EUS Guided Treatment of Gastric Varices
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John DeWitt, Professor of Medicine and Director of Endoscopic Ultrasound, Indiana University
Other Study IDs: 14954
Record Dates: First submitted 2022-08-02; First posted 2022-08-30 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Gastric Varices Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Ultrasound (EUS) administration of cyanoacrylate tissue adhesive to control bleeding gastric varices — Subjects will have undergone treatment and been enrolled into the existing registry.

SUMMARY:
The purpose of the study is to determine the clinical impact of cyanoacrylate tissue adhesive treatment for Gastric Varices performed by Indiana University EUS physicians.

DETAILED DESCRIPTION:
Using an IRB approved database (IU IRB#1209009522; NCT02037659), data collected from the database will be evaluated to identify complications, risk of rebleeding, death within 1 year of treatment, varices eradication and need for re-intervention associated with cyanoacrylate tissue adhesive (Dermabond) treatment performed by Indiana University Endoscopic Ultrasound (EUS) physicians.

ELIGIBILITY:
Inclusion Criteria:

* Any subject enrolled into the existing database (IU IRB#1209009522; NCT02037659).

Exclusion Criteria:

* Not enrolled into the database.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were treated for Gastric Varices with bleeding using cyanoacrylate tissue adhesive and administered by endoscopic ultrasound.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Impact of EUS guided treatment of Gastric varices post procedure complications and adverse events | Complications reviewed at time of retrospective study. EUS-guided sclerotherapy done between November 2012 and December 2021
  Retrospective data review to Determine post procedure complications and adverse events at 24h, between 2 and 7 days and between 8 and 30 days after the procedure. Additionally, tracking rebleeding after first and second EUS. Moreover, looking at eradication of GV rate on second endoscopy (considered eradicated if absent or if residual varices have no or minimal flow on doppler)eradication, and need for re-intervention following cyanoacrylate tissue adhesive treatment for Gastric Varices performed by IU EUS physicians.

CONTACTS AND LOCATIONS:
Overall Officials: John M. DeWitt, MD, Principal Investigator — Professor of Medicine and Director of Endoscopic Ultrasound
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No